CLINICAL TRIAL: NCT07073287
Title: Efficacy of Cerebello-spinal Direct Current Stimulation on Functional Mobility in Chronic Stroke Patients
Brief Title: Efficacy of Cerebello-spinal Direct Current Stimulation (csDCS) on Functional Mobility in Chronic Stroke Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Collaborators: Universidade Federal do Rio de Janeiro (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Kátia Monte-Silva, Professor, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: csDCS_Stroke_Mobility
Record Dates: First submitted 2025-06-18; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Stroke Rehabilitation; Gait Disorders, Neurologic; tDCS
Keywords: spinal cord; stroke; gait; rehabilitation; direct current stimulation
MeSH Terms: conditions — Gait Disorders, Neurologic; Stroke

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial, double blinded (therapist/evaluator, patient) Initial evaluation, followed by 10 days of treatment, followed by a re-evaluation immediately after and follow-up 30 days after finishing.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active cerebello-spinal direct current stimulation (Experimental): csDCS influences both ascending and descending spinal pathways and reflex excitability, promoting prolonged functional neuroplastic changes.
  Interventions: Device: Cerebello-spinal direct current stimulation
- Sham cerebello-spinal direct current stimulation (Sham Comparator): Treadmill training with masking for cerebello-spinal direct current stimulation
  Interventions: Device: Sham Comparator

INTERVENTIONS:
Device: Cerebello-spinal direct current stimulation — csDCS influences both ascending and descending spinal pathways and reflex excitability, promoting prolonged functional neuroplastic changes.
  Other Names: csDCS
  Arms: Active cerebello-spinal direct current stimulation
Device: Sham Comparator — Masking for cerebello-spinal direct current stimulation involves the electric current stopping after 30 seconds, providing a sensation without producing neuromodulation.
  Arms: Sham cerebello-spinal direct current stimulation

SUMMARY:
The aim of this clinical trial is to determine if cerebello-spinal direct current stimulation (csDCS) is effective in treating gait disorders in individuals with chronic stroke. Additionally, the trial seeks to evaluate the safety of this technique.

The primary objectives include:

Investigating whether cerebello-spinal direct current stimulation improves gait and functional mobility in participants with chronic stroke.

Assessing any potential side effects associated with the method.

Researchers will conduct a comparative analysis between cerebello-spinal direct current stimulation and a sham procedure (which mimics the stimulation without any actual effect) to assess its effectiveness in addressing gait disorders and enhancing mobility.

Participants in the trial will:

Undergo cerebello-spinal direct current stimulation combined with treadmill training or a sham procedure with treadmill training daily over a two-week period.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of Stroke by digital or physical imaging or medical report
* Gait impairment
* Stroke with at least 6 months after ictus

Exclusion Criteria:

* Metallic implants in spinal cord
* Major orthopedic/rheumatological disorders
* Inability of verbal or non-verbal communication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Functional Mobility | Baseline, post-treatment (2 weeks) and follow up after 30 days
  The Timed-Up and Go (TUG) test is used to evaluate an individual´s capacity to stand up, walk, and sit down. During the test, the participants are timed from the moment they begin to stand up until they are seated again.

SECONDARY OUTCOMES:
Independency level | Baseline, post-treatment (2 weeks) and follow up after 30 days
  Self-reported independence is assessed using the Functional Ambulation Categories (FAC). Scores range from 0 (inability to walk even with external help) to 5 (normal ambulation).
Lower limb motor function | Baseline, post-treatment (2 weeks) and follow up after 30 days
  Motor function of the lower limbs is assessed using the Fugl-Meyer Assessment, where scores range from 0 (indicating the worst motor function) to 28 (indicating normal motor function).
Balance | Baseline, post-treatment (2 weeks) and follow up after 30 days
  Capacity to maintain balance during various tasks is assessed using the Mini Balance Evaluation System (MiniBEST-test). Its scores range from 0 to 28 points. Lower scores indicate poor balance, while higher scores reflect better balance.
Perceived change in treatment | Upon completion of the two-week intervention
  Evaluation of how the participant describe the perceived change in their condition since the treatment started, using the Patient Global Impression of Change (PGM). This scale assesses the change in activity limitations, symptoms, emotions, and overall quality of life since the beginning of treatment, ranging from no change or worsening to significant improvement that made a considerable difference. A score of one indicates no change, while a score of seven represents a substantial improvement.
Spasticity | Baseline, post-treatment (2 weeks) and follow up after 30 days
  Muscle tone disorders will be assessed using the Modified Ashworth Scale, which measures spasticity by grading muscle resistance during passive stretching. The scale ranges from 0 to 4, where 0 indicates no increase in muscle tone, and 4 represents a limb that is rigid in flexion or extension.

CONTACTS AND LOCATIONS:
Locations (3):
- Brazil (3):
  - Federal University of Paraiba, João Pessoa, Paraíba
  - Federal University of Pernambuco, Recife, Pernambuco
  - Federal University of Rio de Janeiro, Rio de Janeiro, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: Undecided